CLINICAL TRIAL: NCT04223024
Title: Randomized Phase II Trial of Concurrent Chemoradiotherapy With or Without Nimotuzumab for High Risk Nasopharyngeal Carcinoma After Induction Chemotherapy
Brief Title: Concurrent Chemoradiotherapy With Nimotuzumab for High Risk Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2019-191
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCRT + Nimotuzumab (Experimental): Patients whose plasma EBV DNA> 0 copy/mL or SD/PD according to RECIST after two cycle induction chemotherapy( TPF :Paclitaxel liposome135mg/m2 d1+DDP 25mg/m2 d1-d3+ 5-fu 750mg /m2/day civ120h, every 3 weeks for 2 courses) will have concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy) + nimotuzumab (200mg, once a week during radiotherapy, a total of 7 weeks)
  Interventions: Drug: CCRT+Nimotuzumab
- CCRT alone (Active Comparator): Patients whose plasma EBV DNA> 0 copy/mL or SD/PD according to RECIST after two cycle induction chemotherapy( TPF :Paclitaxel liposome135mg/m2 d1+DDP 25mg/m2 d1-d3+ 5-fu 5-fu 750mg /m2/day civ120h, every 3 weeks for 2 courses) will have concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy) )
  Interventions: Drug: CCRT alone

INTERVENTIONS:
Drug: CCRT+Nimotuzumab — concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy) + Nimotuzumab (200mg, once a week during radiotherapy, a total of 7 weeks)
  Other Names: Nimotuzumab
  Arms: CCRT + Nimotuzumab
Drug: CCRT alone — concurrent cisplatin (100mg/m2, every three weeks,D1,D22,D43 of intensity modulated radiotherapy )
  Arms: CCRT alone

SUMMARY:
This is the first phase II randomized clinical trial of concurrent chemoradiotherapy with or without EGFR blocker Nimotuzumab for high risk advanced nasopharyngeal carcinoma(NPC) , determining whether concurrent chemoradiotherapy(CCRT) combined with nimotuzumab can improve the survival rate of high-risk patients and may provide new evidence for individualized comprehensive treatment of locally advanced NPC.

DETAILED DESCRIPTION:
Currently, although NCCN(National Comprehensive Cancer Network) guidelines recommend induction chemotherapy combined with concurrent chemoradiotherapy as IIA level-evidenced treatment for locally advanced nasopharyngeal carcinoma (stage II-IVa),there is still about 20-30% of patients with locally advanced nasopharyngeal carcinoma experienced recurrence and metastasis after radical treatment.

Our previous results showed that patients with plasma Epstein-Barr virus(EBV) DNA> 0 copy/mL or stable disease/progressive disease(SD/PD) after induction chemotherapy had a significantly higher risk of disease progression than patients with plasma EBV DNA=0 copy/mL and complete response/partial response(CR/PR),according to Response Evaluation Criteria in Solid Tumors (RECIST). As for these high-risk patients, the urgent clinical problem to be solved is whether increased treatment intensity during concurrent chemoradiotherapy can improve their survival rates.

Epidermal growth factor (EGFR) is an important therapeutic target for nasopharyngeal carcinoma.Multiple retrospective studies have shown that chemoradiotherapy combined with the EGFR blocker nimotuzumab improved the survival rate of patients with locally advanced nasopharyngeal carcinoma compared with chemoradiotherapy alone. However, phase II randomized clinical trial about the incorporation of nimotuzumab into concurrent chemoradiotherapy is still limited.

This is the first phase II randomized clinical trial of concurrent chemoradiotherapy with or without Nimotuzumab for high risk locally advanced NPC patients, determining whether concurrent chemoradiotherapy combined with nimotuzumab can improve the survival rate of high-risk patients and may provide new evidence for individualized comprehensive treatment of locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, regardless of sex.
2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma with positive EGFR expression, type of WHO II or III, clinical stage II-IVa (according to the 8th American Joint Committee on Cancer[AJCC] edition)
3. Patients with plasma EBV DNA> 0 copy/mL or SD/PD according to RECIST after two cycle induction chemotherapy
4. ECOG (Eastern Cooperative Oncology Group) score: 0-1
5. Women in their reproductive years should ensure that they use contraception during the study period.
6. Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109 /L, platelet (PLT) ≥100×109 /L.
7. Liver function: Alanine transaminase(ALT), Aspartate aminotransferase(AST)< 2.5 times the upper limit of normal value (ULN), total bilirubin <2.0×ULN.
8. Renal function: serum creatinine <1.5×ULN
9. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
2. Receiving radiotherapy or chemotherapy or targeted therapy previously
3. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
4. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
5. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
6. Severe, uncontrolled medical conditions and infections.
7. At the same time using other test drugs or in other clinical trials.
8. Refusal or inability to sign informed consent to participate in the trial.
9. Other treatment contraindications.
10. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) the last follow-up. | 2 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRFS) | 2 years
  Defined from date of randomization to date of first documentation of locoregional relapse or the date of death from any cause or until the date of the last follow-up visit
Distant Metastasis-Free Survival (DMFS) | 2 years
  Defined from date of randomization to date of first documentation of distant metastases or the date of death from any cause or until the date of the last follow-up visit
Objective Response Rate (ORR) | Three months after the completion of the CCRT with or without Nimotuzumab treatment
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI)
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Evaluate EGFR expression level and EGFR Gene Copy Number as a predictive marker for survival outcomes | 2 years
  Pre-treatment EGFR expression level and EGFR Gene Copy Number is evaluated by means of immunohistochemical testing and fluorescent in situ hybridization (FISH), respectively.
Correlation between the frequency of EGFR-specific T cells after treatment and survival outcomes | 2 years
  The frequency of anti-EGFR specific T cells is evaluated centrally by means of flow cytometry
Plasma EBV DNA copy number | 2 years
  Plasma EBV DNA copy number in both arms was assessed by Quantitative real time polymerase chain reaction(qRT-PCR) at pretreatment, after two cycle induction chemotherapy, during CCRT and follow up time . The predictive value of plasma EBV DNA copy number was assessed by survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AW, Lau WH, Tung SY, Chua DT, Chappell R, Xu L, Siu L, Sze WM, Leung TW, Sham JS, Ngan RK, Law SC, Yau TK, Au JS, O'Sullivan B, Pang ES, O SK, Au GK, Lau JT; Hong Kong Nasopharyngeal Cancer Study Group. Preliminary results of a randomized study on therapeutic gain by concurrent chemotherapy for regionally-advanced nasopharyngeal carcinoma: NPC-9901 Trial by the Hong Kong Nasopharyngeal Cancer Study Group. J Clin Oncol. 2005 Oct 1;23(28):6966-75. doi: 10.1200/JCO.2004.00.7542. PMID 16192584
- [Background] Ribassin-Majed L, Marguet S, Lee AWM, Ng WT, Ma J, Chan ATC, Huang PY, Zhu G, Chua DTT, Chen Y, Mai HQ, Kwong DLW, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Bourhis J, Pignon JP, Blanchard P. What Is the Best Treatment of Locally Advanced Nasopharyngeal Carcinoma? An Individual Patient Data Network Meta-Analysis. J Clin Oncol. 2017 Feb 10;35(5):498-505. doi: 10.1200/JCO.2016.67.4119. Epub 2016 Dec 5. PMID 27918720
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Bossi P, Orlandi E, Bergamini C, Locati LD, Granata R, Mirabile A, Parolini D, Franceschini M, Fallai C, Olmi P, Quattrone P, Potepan P, Gloghini A, Miceli R, Mattana F, Scaramellini G, Licitra L. Docetaxel, cisplatin and 5-fluorouracil-based induction chemotherapy followed by intensity-modulated radiotherapy concurrent with cisplatin in locally advanced EBV-related nasopharyngeal cancer. Ann Oncol. 2011 Nov;22(11):2495-2500. doi: 10.1093/annonc/mdq783. Epub 2011 Mar 11. PMID 21398385
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Chan AT, Lo YM, Zee B, Chan LY, Ma BB, Leung SF, Mo F, Lai M, Ho S, Huang DP, Johnson PJ. Plasma Epstein-Barr virus DNA and residual disease after radiotherapy for undifferentiated nasopharyngeal carcinoma. J Natl Cancer Inst. 2002 Nov 6;94(21):1614-9. doi: 10.1093/jnci/94.21.1614. PMID 12419787
- [Background] Hou X, Zhao C, Guo Y, Han F, Lu LX, Wu SX, Li S, Huang PY, Huang H, Zhang L. Different clinical significance of pre- and post-treatment plasma Epstein-Barr virus DNA load in nasopharyngeal carcinoma treated with radiotherapy. Clin Oncol (R Coll Radiol). 2011 Mar;23(2):128-33. doi: 10.1016/j.clon.2010.09.001. Epub 2010 Oct 12. PMID 20943358
- [Background] Liu LT, Tang LQ, Chen QY, Zhang L, Guo SS, Guo L, Mo HY, Zhao C, Guo X, Cao KJ, Qian CN, Zeng MS, Bei JX, Hong MH, Shao JY, Sun Y, Ma J, Mai HQ. The Prognostic Value of Plasma Epstein-Barr Viral DNA and Tumor Response to Neoadjuvant Chemotherapy in Advanced-Stage Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2015 Nov 15;93(4):862-9. doi: 10.1016/j.ijrobp.2015.08.003. Epub 2015 Aug 7. PMID 26530755
- [Background] Huang CL, Sun ZQ, Guo R, Liu X, Mao YP, Peng H, Tian L, Lin AH, Li L, Shao JY, Sun Y, Ma J, Tang LL. Plasma Epstein-Barr Virus DNA Load After Induction Chemotherapy Predicts Outcome in Locoregionally Advanced Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):355-361. doi: 10.1016/j.ijrobp.2019.01.007. Epub 2019 Jan 23. PMID 30682489
- [Background] Ciardiello F, Tortora G. A novel approach in the treatment of cancer: targeting the epidermal growth factor receptor. Clin Cancer Res. 2001 Oct;7(10):2958-70. PMID 11595683
- [Background] Mendelsohn J. Targeting the epidermal growth factor receptor for cancer therapy. J Clin Oncol. 2002 Sep 15;20(18 Suppl):1S-13S. No abstract available. PMID 12235219
- [Background] Chua DT, Nicholls JM, Sham JS, Au GK. Prognostic value of epidermal growth factor receptor expression in patients with advanced stage nasopharyngeal carcinoma treated with induction chemotherapy and radiotherapy. Int J Radiat Oncol Biol Phys. 2004 May 1;59(1):11-20. doi: 10.1016/j.ijrobp.2003.10.038. PMID 15093894
- [Background] Ramakrishnan MS, Eswaraiah A, Crombet T, Piedra P, Saurez G, Iyer H, Arvind AS. Nimotuzumab, a promising therapeutic monoclonal for treatment of tumors of epithelial origin. MAbs. 2009 Jan-Feb;1(1):41-8. doi: 10.4161/mabs.1.1.7509. PMID 20046573
- [Background] Huang JF, Zhang FZ, Zou QZ, Zhou LY, Yang B, Chu JJ, Yu JH, Zhang HW, Yuan XP, Tai GM, Liu FJ, Ma CC. Induction chemotherapy followed by concurrent chemoradiation and nimotuzumab for locoregionally advanced nasopharyngeal carcinoma: preliminary results from a phase II clinical trial. Oncotarget. 2017 Jan 10;8(2):2457-2465. doi: 10.18632/oncotarget.13899. PMID 27974693
- [Background] Wang F, Sun Q, Jiang C, Liu T, Rihito A, Masoto S, Wang Y, Fu Z, Chen M. Additional induction chemotherapy to concurrent chemotherapy and intensity-modulated radiotherapy with or without nimotuzumab in first-line treatment for locoregionally advanced nasopharyngeal carcinoma: a propensity score matched analysis. J Cancer. 2018 Jan 1;9(3):594-603. doi: 10.7150/jca.20461. eCollection 2018. PMID 29483965
- [Background] Liu ZG, Zhao Y, Tang J, Zhou YJ, Yang WJ, Qiu YF, Wang H. Nimotuzumab combined with concurrent chemoradiotherapy in locally advanced nasopharyngeal carcinoma: a retrospective analysis. Oncotarget. 2016 Apr 26;7(17):24429-35. doi: 10.18632/oncotarget.8225. PMID 27016412
- [Background] Fangzheng W, Chuner J, Zhiming Y, Tongxin L, Fengqin Y, Lei W, Bin L, Fujun H, Ming C, Weifeng Q, Zhenfu F. Long-Term Use of Nimotuzumab in Combination With Intensity-Modulated Radiotherapy and Chemotherapy in the Treatment of Locoregionally Advanced Nasopharyngeal Carcinoma: Experience of a Single Institution. Oncol Res. 2018 Mar 5;26(2):277-287. doi: 10.3727/096504017X15079846743590. Epub 2017 Oct 18. PMID 29046165